CLINICAL TRIAL: NCT06070480
Title: Effects of Propofol, Desflurane and Spinal Anesthesia on Intraocular Pressure During Lumbar Disc Herniation Surgery: A Randomized Controlled Study
Brief Title: Effects of Different Types of Anaesthesia on Intraocular Pressure During Lumbar Disc Herniation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Elvan Yilmaz, Assistant professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KAEK 04/2020
Record Dates: First submitted 2023-09-18; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia; Disk Herniated Lumbar; Intraocular Pressure
Keywords: prone position; intraocular pressure; hemodynamics; anesthesia,spinal; anesthesia,general

STUDY DESIGN:
Intervention Model Description: The study included 75 patients with lumbar disc herniation between the ages of 18-75, with the American Society of Anesthesiologists (ASA) 1-2. The patients were randomly divided into 3 groups: propofol, desflurane, spinal. Intraocular pressure was measured at 5 time points throughout surgery, including baseline (T1), 10 minutes after anesthesia (T2), 10 minutes after prone positioning (T3: early prone), 30 minutes after prone positioning (T4: late prone), and 10 minutes after returning to the supine position (T5). Hemodynamic parameters were measured at these time points. Hemoglobin and hematocrit values were measured preoperatively and on the first postoperative day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal Anesthesia Group (Active Comparator): Intraocular pressure values of the patients operated with spinal anaesthesia were measured
  Interventions: Other: Spinal Anesthesia Group
- Desflurane Group (Active Comparator): Intraocular pressure values were measured in patients operated under general anaesthesia with desflurane.
  Interventions: Other: Desflurane Group
- Propofol Group (Active Comparator): Intraocular pressure values were measured in patients operated under general anaesthesia with desflurane.
  Interventions: Other: Propofol Group

INTERVENTIONS:
Other: Spinal Anesthesia Group — Effect of spinal anesthesia on intraocular pressure
  Arms: Spinal Anesthesia Group
Other: Desflurane Group — Effect of general anesthesia with desflurane on intraocular pressure
  Arms: Desflurane Group
Other: Propofol Group — Effect of general anesthesia with propofol on intraocular pressure
  Arms: Propofol Group

SUMMARY:
The aim of this study was to investigate the effects of anaesthesia methods on intraocular pressure during lumbar disc surgery performed in the prone position.

DETAILED DESCRIPTION:
The study included 75 patients with lumbar disc herniation between the ages of 18-75, with the American Society of Anesthesiologists (ASA) 1-2. The patients were randomly divided into 3 groups: propofol, desflurane, spinal. Intraocular pressure (IOP) was measured at 5 time points throughout surgery, including baseline (T1), 10 minutes after anesthesia (T2), 10 minutes after prone positioning (T3: early prone), 30 minutes after prone positioning (T4: late prone), and 10 minutes after returning to the supine position (T5). Hemodynamic parameters were measured at these time points. Hemoglobin and hematocrit values were measured preoperatively and on the first postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 according to the American Society of Anesthesiologists (ASA) Classification.

Exclusion Criteria:

* Who did not sign the informed consent form,
* patients who required emergency surgery,
* eye surgery recipients,
* subjects with acute or chronic eye diseases other than refractive errors,
* individuals detected to have elevated IOP in preoperative measurements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | Time 1:baseline supine , Time 2: 10. minute supine, Time 3: 20. minute prone , Time 4: 30. minute prone,Time 5: 10. minute after returning to the supine
  Intraocular pressure was measured a total of 5 times at set time points throughout the procedures.

SECONDARY OUTCOMES:
Mean Arterial Pressure | Time 1:baseline supine , Time 2: 10. minute supine, Time 3: 20. minute prone , Time 4: 30. minute prone,Time 5: 10. minute after returning to the supine
  Mean Arterial Pressure was measured a total of 5 times at set time points throughout the procedures.
Heart Rate | Time 1:baseline supine , Time 2: 10. minute supine, Time 3: 20. minute prone , Time 4: 30. minute prone,Time 5: 10. minute after returning to the supine
  Heart Rate was measured a total of 5 times at set time points throughout the procedures.
End Tidal Carbon Dioxide (CO2) | Time 1:baseline supine , Time 2: 10. minute supine, Time 3: 20. minute prone , Time 4: 30. minute prone,Time 5: 10. minute after returning to the supine
  End Tidal CO2 was measured a total of 5 times at set time points throughout the procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Elvan Tekir Yılmaz, M.D., Principal Investigator — Giresun University
Locations (1):
- Elvan Tekir Yılmaz, Giresun, Gi̇resun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunha PD, Barbosa TP, Correia G, Silva R, Cruz Oliveira N, Varanda P, Direito-Santos B. The ideal patient positioning in spine surgery: a preventive strategy. EFORT Open Rev. 2023 Feb 21;8(2):63-72. doi: 10.1530/EOR-22-0135. PMID 36805330
- [Result] Kwee MM, Ho YH, Rozen WM. The prone position during surgery and its complications: a systematic review and evidence-based guidelines. Int Surg. 2015 Feb;100(2):292-303. doi: 10.9738/INTSURG-D-13-00256.1. PMID 25692433
- [Result] DePasse JM, Palumbo MA, Haque M, Eberson CP, Daniels AH. Complications associated with prone positioning in elective spinal surgery. World J Orthop. 2015 Apr 18;6(3):351-9. doi: 10.5312/wjo.v6.i3.351. eCollection 2015 Apr 18. PMID 25893178
- [Result] Pinar HU, Kasdogan ZEA, Basaran B, Coven I, Karaca O, Dogan R. The effect of spinal versus general anesthesia on intraocular pressure in lumbar disc surgery in the prone position: A randomized, controlled clinical trial. J Clin Anesth. 2018 May;46:54-58. doi: 10.1016/j.jclinane.2018.01.026. Epub 2018 Mar 26. PMID 29414618
- [Derived] Yilmaz ET, Keles BO. Effects of propofol, desflurane, and spinal anesthesia on intraocular pressure during lumbar disc herniation surgery: a randomized controlled study. Eur Rev Med Pharmacol Sci. 2024 Feb;28(4):1407-1416. doi: 10.26355/eurrev_202402_35462. PMID 38436174